CLINICAL TRIAL: NCT06119724
Title: Bipolar Enbloc Versus Thulium-Yag Enbloc Resection Of Bladder Tumors: A Randomized Controlled Trial
Brief Title: Bipolar Enbloc Versus Thulium-Yag Enbloc Resection of Bladder Tumors
Acronym: TURBT-Enbloc
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Omar, Associate professor of urology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bipolar and Thulium-Yag Enbloc
Record Dates: First submitted 2023-06-17; First posted 2023-11-07 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar enbloc resection of bladder tumors (Active Comparator): Patients who have odd number will be in the first group which will be enrolled in bipolar enbloc group
  Interventions: Procedure: Bipolar enbloc resection of bladder tumor
- Thulium enbloc resection of bladder tumors (Active Comparator): patients who have even number will be in the second group which will be Thulium-Yag laser enbloc group
  Interventions: Procedure: Thulium laser enbloc resection of bladder tumor

INTERVENTIONS:
Procedure: Bipolar enbloc resection of bladder tumor — Enbloc retrival of bladder tumor entoto using cystoscopy using bipolar
  Arms: Bipolar enbloc resection of bladder tumors
Procedure: Thulium laser enbloc resection of bladder tumor — Enbloc retrival of bladder tumor entoto using cystoscopy using thulium laser
  Arms: Thulium enbloc resection of bladder tumors

SUMMARY:
Prospective controlled study randomized comparing bipolar enbloc versus thulium enbloc for bladder tumours

DETAILED DESCRIPTION:
Bladder cancer is the ninth most prevalent cancer worldwide and the 2nd most common urologic cancer in the last two decades after cancer prostate .

Most bladder cancers attributed to exposure to environmental and occupational chemicals, the largest of which by far is tobacco smoke. Greater tobacco smoke and occupational exposure in men may help in the explanation of the 4-fold gender difference in bladder cancer incidence .

Approximately 75-85% of patients with bladder cancer present with disease confined to the mucosa or submucosa , which is referred to as nonmuscle invasive bladder cancer (NMIBC).

Transurethral resection of bladder tumor (TURBT) is still considered the gold standard treatment for primary nonmuscle invasive bladder cancer.

There are many drawbacks for conventional TURBT procedure such as such as the deficiency of the bladder detrusor muscle In the specimen

, the obturator jerk, thermal damage to surrounding tissues, and the technique of( incise and scatter). These drawbacks may lead to difficulty in performing an accurate pathological evaluation of fragment tissue and increase the risk of recurrence.

Laser therapy for bladder cancer was first reported in Germany in the 1970s and was approved to clinical use in the USA in 1984.

Modern laser technology has led to new alternatives to conventional transurethral resection of bladder tumor (TURBT) due to its efficacy and good control of bleeding. With the introduction of en-bloc resection of urinary bladder tumors, Laser come back into focus. The two most commonly used lasers at present are thulium and holmium Laser.

In 2018 PA Geavlete, declared that the enbloc bipolar resection of bladder tumors using mushroom loop provide the advantages of superior surgical safety, decreased perioperative morbidity and faster postoperative recovery, when compared to the standard monopolar TURBT but showed no superiority in oncological outcome.

ELIGIBILITY:
* Inclusion criteria:

  1. Patients with NMIBC
  2. Bladder tumors<4 cm in CT.
  3. Resectable bladder tumors.
  4. Age <80 years.
* Exclusion criteria :

  1. Bladder tumours > 4cm .
  2. Metastatic bladder tumors.
  3. Patients with carcinoma in situ CIS .
  4. Patients with coagulopathies.
  5. Domal bladder tumors.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-11 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Enbloc technique effectiveness in obtaining muscle in the speciment | 3 months
  Assessed by presence of muscles in histopathological specimen.
Duration of cancer free survival post enbloc resection | 1year
  Duration of Cancer free survival post resection measured by weeks.
Staging of bladder cancer post enbloc resection | 1year
  Clinical staging using bimanual examination under anesthesia.
Presence of residual tumors post resection | 3-6 months
  Assessed by visualization of any residual mass during second look cystoscopy
Blood loss | Immediate postoperative
  Assessed by comparing between Hemoglobin level pre and post operative

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia university hospital, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Yes